CLINICAL TRIAL: NCT05950295
Title: Intranasal Lavage With Hypochlorous Acid Safely Reduces the Symptoms in the Ambulatory Patient With COVID-19.
Status: Completed | Type: Observational
Sponsor: Monique Lisa Abner (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 036-020
Record Dates: First submitted 2023-07-15; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
Keywords: intranasal lavage
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Intranasal lavage with hypochlorous acid solution — intranasal lavage for ten days

SUMMARY:
The goal of this observational study is to determine if intranasal lavage reduces symptoms in adults with COVID-19. The main question is can a hypochlorous acid solution reduce the symptoms of COVID-19.

Participants will asked to do the following:

* Irrigate each nostril once a day for ten days with a hypochlorous acid solution.
* Write a daily record of the presence or absence of symptoms such as fever, headache, chills, nausea, or change in sense of smell.
* After ten days, return the daily log in the mail to the investigator.

DETAILED DESCRIPTION:
Methods This study was approved by the Institutional Review Board of Reading Hospital (IRB 036-020) with informed consent obtained from all adult participants. Convenience sampling methodology was utilized for those who met the study criteria inclusive to all gender at ages18 years old and/or older. Excluded participants were those who expressed the desire to not use nasal lavage, women with known pregnancies, and children aged 17 years old and/or younger. The source of enrollees was generated from patients presenting to an ambulatory testing facility for nasopharyngeal swabs for COVID-19. Swab analysis was obtained by reverse transcription-polymerase chain reaction until the COVID-19 antigen specific test (Binax NOW, Abbott Lab) became available for use which allowed a more lenient process for including the Covid-19 positive patients. Each enrolled participant was given a Nasaflo Neti Pot (NeilMed Pharmaceuticals, Inc) with instructions to irrigate each nostril once a day for ten days with the provided hypochlorous solution Vashe Wound Solution (Urgo Medical North America, LLC). Each participant began the daily 120 cc (four -ounce) nasal lavage intervention within 72 hours of their testing. Each participant was given a scripted diary log in which they recorded daily the presence or absence of clinical symptoms such as elevated temperature, fatigue, headache, chills, nausea, and anosmia by noting "yes" or "no." After completing the ten days of nasal lavage, each log was returned to the principal investigator via mail. The participants remained quarantined for the recommended time period of 14 days, and adhered to social distancing, handwashing, and donning of face masks. Throughout the study, each participant was urged to not share their devices with any other individuals. After thirty days from the start of their nasal intervention, participants were telephoned for a follow-up review.

ELIGIBILITY:
Inclusion Criteria:

* All gender aged 18 years and older.
* Positive COVID-19 specific antigen test resulted within 72 hours.

Exclusion Criteria:

* Persons with known current pregnancy
* Persons less than or equal to 17 years of age.
* Persons currently using any intranasal medications or agents
* Persons unwilling to use nasal lavage.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The source of enrollees was generated from persons presenting to one ambulatory testing facility for nasopharyngeal swab testing for COVID-19.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-03-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Reduction in symptoms of COVID-19 | 40 days from start of nasal lavage
  Change in sense of smell, fever profile, nasal congestion, and headache

CONTACTS AND LOCATIONS:
Locations (1):
- Tower Health/Reading Hospital, Reading, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joynt GM, Wu WK. Understanding COVID-19: what does viral RNA load really mean? Lancet Infect Dis. 2020 Jun;20(6):635-636. doi: 10.1016/S1473-3099(20)30237-1. Epub 2020 Mar 27. No abstract available. PMID 32224308
- [Background] Waradon S, Ni H, Christophe B, Marjjin B. SARS-CoV-2 Entry Genes Are Most Highly Expressed in Nasal Goblet and Ciliated Cells Within Human Airway.Nature Medicine. 2020. Mar.arXiv.org.
- [Background] Wang L, Bassiri M, Najafi R, Najafi K, Yang J, Khosrovi B, Hwong W, Barati E, Belisle B, Celeri C, Robson MC. Hypochlorous acid as a potential wound care agent: part I. Stabilized hypochlorous acid: a component of the inorganic armamentarium of innate immunity. J Burns Wounds. 2007 Apr 11;6:e5. PMID 17492050
- [Background] Robson MC, Payne WG, Ko F, Mentis M, Donati G, Shafii SM, Culverhouse S, Wang L, Khosrovi B, Najafi R, Cooper DM, Bassiri M. Hypochlorous Acid as a Potential Wound Care Agent: Part II. Stabilized Hypochlorous Acid: Its Role in Decreasing Tissue Bacterial Bioburden and Overcoming the Inhibition of Infection on Wound Healing. J Burns Wounds. 2007 Apr 11;6:e6. PMID 17492051
- [Background] Stroman DW, Mintun K, Epstein AB, Brimer CM, Patel CR, Branch JD, Najafi-Tagol K. Reduction in bacterial load using hypochlorous acid hygiene solution on ocular skin. Clin Ophthalmol. 2017 Apr 13;11:707-714. doi: 10.2147/OPTH.S132851. eCollection 2017. PMID 28458509
- [Background] Farrell NF, Klatt-Cromwell C, Schneider JS. Benefits and Safety of Nasal Saline Irrigations in a Pandemic-Washing COVID-19 Away. JAMA Otolaryngol Head Neck Surg. 2020 Sep 1;146(9):787-788. doi: 10.1001/jamaoto.2020.1622. No abstract available. PMID 32722777
- [Background] Ramalingam S, Graham C, Dove J, Morrice L, Sheikh A. A pilot, open labelled, randomised controlled trial of hypertonic saline nasal irrigation and gargling for the common cold. Sci Rep. 2019 Jan 31;9(1):1015. doi: 10.1038/s41598-018-37703-3. PMID 30705369
- [Background] Guenezan J, Garcia M, Strasters D, Jousselin C, Leveque N, Frasca D, Mimoz O. Povidone Iodine Mouthwash, Gargle, and Nasal Spray to Reduce Nasopharyngeal Viral Load in Patients With COVID-19: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Apr 1;147(4):400-401. doi: 10.1001/jamaoto.2020.5490. PMID 33538761
- [Background] Hakim H, Thammakarn C, Suguro A, Ishida Y, Kawamura A, Tamura M, Satoh K, Tsujimura M, Hasegawa T, Takehara K. Evaluation of sprayed hypochlorous acid solutions for their virucidal activity against avian influenza virus through in vitro experiments. J Vet Med Sci. 2015 Feb;77(2):211-5. doi: 10.1292/jvms.14-0413. Epub 2014 Nov 24. PMID 25421399
- [Background] Ramalingam S, Cai B, Wong J, Twomey M, Chen R, Fu RM, Boote T, McCaughan H, Griffiths SJ, Haas JG. Antiviral innate immune response in non-myeloid cells is augmented by chloride ions via an increase in intracellular hypochlorous acid levels. Sci Rep. 2018 Sep 11;8(1):13630. doi: 10.1038/s41598-018-31936-y. PMID 30206371
- [Background] Wang G. Chloride flux in phagocytes. Immunol Rev. 2016 Sep;273(1):219-31. doi: 10.1111/imr.12438. PMID 27558337
- [Result] Spinato G, Fabbris C, Polesel J, Cazzador D, Borsetto D, Hopkins C, Boscolo-Rizzo P. Alterations in Smell or Taste in Mildly Symptomatic Outpatients With SARS-CoV-2 Infection. JAMA. 2020 May 26;323(20):2089-2090. doi: 10.1001/jama.2020.6771. PMID 32320008